CLINICAL TRIAL: NCT00997347
Title: The Extended Gestational Age Medical Abortion Study: The Effectiveness of Medical Abortion With Mifepristone and Misoprostol at 57-63 Days Versus 64-70 Days Gestation
Brief Title: The Extended Gestational Age Medical Abortion Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1.2.2
Record Dates: First submitted 2009-10-01; First posted 2009-10-19 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Medical Abortion
MeSH Terms: interventions — Mifepristone; Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 64-70 days' gestational age (Experimental): Women whose pregnancies are estimated to have a gestational age of 64-70 days
  Interventions: Drug: Mifepristone and misoprostol
- 57-63 days' gestational age (No Intervention): Women whose pregnancies are estimated to have a gestational age of 57-63 days. (Women in this arm receive the standard of care for medical termination of pregnancy in the stated gestational age range.)

INTERVENTIONS:
Drug: Mifepristone and misoprostol — 200 mg oral mifepristone
  800 mcg buccal misoprostol or 400 mcg sublingual misoprostol 24-48 hours after mifepristone
  Arms: 64-70 days' gestational age

SUMMARY:
This open-label, comparative study will compare the efficacy, safety, and acceptability of 200 mg mifepristone followed in 24-48 hours by 800mcg buccal misoprostol or 400mcg sublingual misoprostol for termination of pregnancy in existing outpatient early medical abortion services among women 57-63 days' versus 64-70 days' gestation.

ELIGIBILITY:
Inclusion Criteria:

* intrauterine pregnancy of greater than 56 days and less than 71 days
* eligible for medical abortion according to study doctor assessment
* willing and able to sign consent forms
* speak English or Spanish (in US sites); speak the local language(s) (in international sites)
* agree to comply with the study procedures and visit schedule

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1400 (Actual)
Dates: Start 2009-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Efficacy: Proportion of women who successfully complete abortion without surgical intervention to resolve viable pregnancy or incomplete abortion | 7-36 days

SECONDARY OUTCOMES:
Proportion of individual side effects experienced by participants | 7-14 days
Proportion of women who determined method acceptable (i.e., overall acceptability of method, time to abortion completion, bleeding, side effects, and pain) | 7-14 days
Bleeding patterns, i.e. proportion of women who experienced heavy, moderate, or light bleeding according by day since abortion began | 7-14 days
Average number of missed days of work or school due to the abortion procedure | 7-14 days

CONTACTS AND LOCATIONS:
Overall Officials: Yael Swica, MD, MPH, Principal Investigator — Gynuity Health Projects; Hillary Bracken, PhD, Principal Investigator — Gynuity Health Projects; Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects
Locations (12):
- United States (6):
  - Presidential Women's Center, West Palm Beach, Florida
  - Family Planning Associates Medical Group, Chicago, Illinois
  - Planned Parenthood League of Massachusetts, Boston, Massachusetts
  - Planned Parenthood, Minnesota, North Dakota, South Dakota, Saint Paul, Minnesota
  - Planned Parenthood of New York City, New York, New York
  - Planned Parenthood, Central Texas, Waco, Texas
- Zhordania Institute of Human Reproduction, Tbilisi, Georgia
- India (2):
  - Government Medical College (GMC), Nagpur
  - Naval Nursing Home, Solapur
- La Rabta Maternity Hospital, Tunis, Tunisia
- Ukraine (2):
  - Central District Maternity House, Odesa
  - Maternity Hospital No.2, Simferopol

REFERENCES:
- [Derived] Winikoff B, Dzuba IG, Chong E, Goldberg AB, Lichtenberg ES, Ball C, Dean G, Sacks D, Crowden WA, Swica Y. Extending outpatient medical abortion services through 70 days of gestational age. Obstet Gynecol. 2012 Nov;120(5):1070-6. doi: 10.1097/aog.0b013e31826c315f. PMID 23090524